CLINICAL TRIAL: NCT04488926
Title: Efficacy and Tolerability of Micronized and Ultramicronized Palmitoylethanolamide in Fibromyalgia Patients: A Double-blind, Randomized, Placebo-controlled Clinical Trial
Brief Title: Micronized and Ultramicronized Palmitoylethanolamide in Fibromyalgia Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Epitech Group SpA (Industry)
Collaborators: Azienda Ospedaliera Universitaria Integrata Verona (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: MPS-FM
Record Dates: First submitted 2020-07-20; First posted 2020-07-28 (Actual); Last update posted 2023-09-07 (Actual); Status verified 2023-02

CONDITIONS: Fibromyalgia
MeSH Terms: conditions — Fibromyalgia | interventions — Standard of Care; Drug Repositioning; Acetaminophen

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1 (Active Comparator): Normast® MPS (mPEA and umPEA 300mg + 600mg) microgranules for sublingual use, 1800mg/die in 2 doses (morning and evening) for 90 days
  Interventions: Dietary Supplement: micronized and ultra-micronized Palmitoylethanolamide (mPEA and umPEA, 300mg + 600mg) microgranules; Drug: Standard Therapy; Drug: Rescue Drug
- Group 2 (Placebo Comparator): Placebo microgranules for sublingual use, 1800mg/die in 2 doses (morning and evening) for 90 days
  Interventions: Other: Placebo microgranules 1800mg; Drug: Standard Therapy; Drug: Rescue Drug

INTERVENTIONS:
Dietary Supplement: micronized and ultra-micronized Palmitoylethanolamide (mPEA and umPEA, 300mg + 600mg) microgranules — Micronized and ultra-micronized Palmitoylethanolamide is on the market in Italy as a Food for Special Medical Purposes
  Other Names: Normast® MPS microgranules
  Arms: Group 1
Other: Placebo microgranules 1800mg — Placebo was prepared to be indistinguishable from color and flavor from the Product
  Arms: Group 2
Drug: Standard Therapy — (antidepressants, anticonvulsants, muscle relaxants, weak opiates, etc..) consolidated for at least 3 months
Drug: Rescue Drug — Use as needed allowed
  Other Names: Paracetamol or Fans

SUMMARY:
The onset of chronic Fibromyalgia symptomatology is due to central alterations, together with peripheral neuroimmune modifications. Using positron emission tomography (PET), it has been observed for the first time that fibromyalgia patients have a high activation of microglial cells compared to normal subjects. Experimental evidence in neuroinflammation models in vitro and in vivo have demonstrated the anti-inflammatory and neuroprotective effect of Palmitoylethanolamide (PEA), effects confirmed by observational clinical investigations conducted in patients with fibromyalgia in which micronized and ultra-micronized Palmitoylethanolamide (mPEA and umPEA) reduced the intensity of pain improving the quality of life. The aim of this study is to investigate the efficacy and tolerability of PEA-m + PEA-um administered as an add-on therapy with a double-blind, randomized, placebo-controlled clinical investigation.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Fibromyalgia according to the criteria of the American College of Rheumatology 2016 (symptoms for at least 3 months, Widespread Pain Index (WPI) ≥ 7 and Symptom Severity (SS) ≥ 5 or WPI 4-6 and SS ≥ 9)
* Pain intensity assessed on the Visual Analogue Scale (VAS) ≥ 40
* PEA-naive patients
* Patients who agree to sign informed consent

Exclusion Criteria:

* Values of WPI <7 and SS <5
* Pain intensity assessed on the Visual Analogue Scale (VAS) <40
* Patients who have already taken PEA in the past
* Allergic or hypersensitive subjects to the product and / or one or more of its excipients
* Patients who refuse to sign informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2020-07-16 (Actual); Primary Completion 2022-05-02 (Actual); Study Completion 2022-05-02 (Actual)

PRIMARY OUTCOMES:
Fibromyalgia symptoms assessed by Fibromyalgia Impact Questionnaire Revised | 90 days
  Change of Fibromyalgia symptoms

SECONDARY OUTCOMES:
Pain Intensity assessed by Visual Analogue Scale | 90 days
  Change of Visual Analogue Scale every 30 days (0: no pain - 100 mm: maximum pain)
Health assessed by Short form-12 Health Survey | 90 days
  Change in Health at the end of treatment
Sleep Disorders assessed by Pittsburgh Sleep Quality Index | 90 days
  Change in sleep disorders at the end of treatment
Rescue Drugs consumption assessed by a daily diary | 90 days
  Change in rescue drugs consumption during the entire period
Incidence of Adverse Events | 90 days
  Monitoring of adverse event
Blood test | 90 days
  Clinically significant changes in blood test

CONTACTS AND LOCATIONS:
Overall Officials: Enrico Polati, MD, Principal Investigator — Azienda Ospedaliera Universitaria Integrata di Verona
Locations (1):
- Anestesia e Rianimazione B - Azienda Ospedaliera Universitaria Integrata di Verona, Verona, VR, Italy

REFERENCES:
- [Background] Schweiger V, Martini A, Bellamoli P, Donadello K, Schievano C, Balzo GD, Sarzi-Puttini P, Parolini M, Polati E. Ultramicronized Palmitoylethanolamide (um-PEA) as Add-on Treatment in Fibromyalgia Syndrome (FMS): Retrospective Observational Study on 407 Patients. CNS Neurol Disord Drug Targets. 2019;18(4):326-333. doi: 10.2174/1871527318666190227205359. PMID 30827269
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/30827269/